CLINICAL TRIAL: NCT01594164
Title: Clinical Study to Assess Change in Upper Airway Geometry Between Upright and Supine Position
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FLUIDDA nv (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: FLUI-2010-61
Record Dates: First submitted 2012-05-03; First posted 2012-05-08 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Changes in Upper Airway Geometry
Keywords: High Resolution Computed Tomography; Cone Beam Computed Tomography; upper airway; geometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Cone Beam Computed Tomography — CBCT scan of upper airway, in upright position.
  Other Names: CBCT
Radiation: High Resolution Computed Tomography — HRCT scan of upper airway, in supine position.
  Other Names: HRCT

SUMMARY:
In this study the changes in upper airway geometry and resistance between images, obtained in upright and supine position, will be evaluated. Therefore a Cone Beam Computed Tomography (CBCT) scan and a low dose Computed Tomography (CT) scan will be taken in a population of 20 subjects. The upright morphology will be obtained using CBCT scan while the supine upper airway geometry will be determined using a standard High Resolution Computed Tomography (HRCT) scanner.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained.
* Male or female subject aged ≥ 18 years.
* BMI < 25 kg/m2 (group 1), BMI ≥ 25 kg/m2 and < 30 kg/m2 (group 2) and BMI ≥ 30 kg/m2 (group 3) at visit 0. BMI calculation should be repeated if the interval visit 0 - visit 1 > 14 days.
* Female subject of childbearing potential who confirms that a contraception method was used at least two months before visit 1.

Exclusion Criteria:

* Subject is under the age of legal consent.
* Subject who is pregnant or is breast-feeding.
* Subject with a history of surgery of the upper airway.
* Subject with a history of any illness that, in opinion of the investigator, might confound the results of the study or poses an additional risk to the subject by participation in the study.
* Subject is unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study.
* Subject who received any investigational new drug within the last 4 weeks prior to visit 1.
* Subject who has claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Changes in upper airway geometry | At day 1
  The primary objective of this study is to compare the volume and resistance of the upper airway in supine versus upright position using High Resolution Computed Tomography (HRCT) and Cone Beam Computed Tomography (CBCT) images.

SECONDARY OUTCOMES:
Body mass index (BMI) | At screening and also at day 1 (if interval screening - day 1 > 14 days)
  In addition the effect of elevated BMI on the changes in upper airway morphology will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Backer, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium